CLINICAL TRIAL: NCT00278603
Title: Hematopoietic Stem Cell Injection for Peripheral Vascular Disease: Induction of Neoangiogenesis. A Phase I Study
Brief Title: Stem Cell Injection for Peripheral Vascular Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVD.HSCT2003
Record Dates: First submitted 2006-01-15; First posted 2006-01-18 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Stem Cell Transplantation — Autologous Hematopoietic Stem Cell Injection

SUMMARY:
Severe peripheral vascular disease of the legs causes narrowing of the blood vessels in the legs, which keeps the blood from flowing adequately through these vessels. This study is designed to examine whether treating patients with their own previously collected blood stem cells will improve blood flow in the most severely affected leg. Blood stem cells are undeveloped cells that have the capacity to grow into mature blood cells, which normally circulate in the blood stream.

ELIGIBILITY:
Inclusion Criteria:

* Atherosclerotic ischemic peripheral vascular disease with rest pain defined as pain that occurs at night or at rest that involves the foot and is a sign of end stage vascular disease and / or ischemic lower extremity ulcers due to infra-inguinal disease and/or peak walking time of 1 to 6 minutes on two exercise tests separated by 2 weeks on graded treadmill.
* Either a or b

  1. Ankle brachial index (ABI) < 1.0.
  2. Doppler waveforms at posterior tibial artery and dorsalis pedis artery are monophasic with toe pressure < 30 mmHg.
* A non-surgical candidate for revascularization e.g. prior vascular reconstruction, inability to locate a suitable vein for grafting, diffuse multi- segment disease, or extensive infra-popliteal disease not amenable to a vascular graft.
* Age > 18 years old.

Exclusion Criteria:

* Popliteal vascular entrapment syndrome
* Lower Extremity infection or infected ulcer
* Hypercoagulable state
* HIV positive
* HBsAg positive
* Uncontrolled arrhythmia, that is, persistence of an arrhythmia despite medical therapy
* Unstable angina
* Thrombocytopenia < 100,000/ul
* Anemia that cannot be transfused to a hemoglobin greater than 10 g/dl
* Leukemia or myelodysplasia
* Allergy to E coli or its products
* Patients with metal in their bodies cannot undergo MRIs (MRA). Therefore, patients with, cochlear implants, or aneurysm clips are not eligible. Coronary artery stents are not a contraindication. Patients with pacemakers are still candidates provided they have normal creatinine (< 1.1 mg/dl) and can receive contrast dye (no allergy) for angiogram instead of MRA.
* Patients who are pregnant
* Poorly controlled diabetes (HbA1c > 6.5)
* Current malignancy, except squamous cell or basal cell skin cancers thought to be easily controlled.
* AST, ALT, or bilirubin more than twice the upper limit of normal.
* WBC < 2.5 / ul.
* Any patient who is actively bleeding, including blood on urine dipstick or fecal occult blood.
* No patient may be re-treated until at least 5 patients have completed 6 months of follow-up with no notable safety findings and evidence of therapeutic efficacy (improved ABI or healing ulcer) occurred at stem cell doses higher than the patient received in this dose escalation study or response occurred in the treated leg and the untreated leg meets eligibility criteria. Re-treated patients must meet eligibility criteria.
* Patients who smoke unless stop smoking at least two weeks before enrollment and agree not to smoke thereafter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The Primary outcome is safety. Safety parameters are survival, and complications related to therapy such as bleeding, infection, acute thrombus or calcification. | 2 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: William Pearce, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States